CLINICAL TRIAL: NCT04992793
Title: Paediatric Brain Injury Following Cardiac Interventions (BICI 2 Kids Study)
Brief Title: Paediatric Brain Injury Following Cardiac Interventions
Acronym: BICI2Kids
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0777
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Congenital heart surgery — Paediatric congenital heart surgery

SUMMARY:
Children born with congenital heart problems face numerous physical, developmental, and social challenges. Complications in pregnancy have potential to impair brain development, leading a smaller brain volume and less mature brain even in babies born at full term. As the brain is less mature, it may be more susceptible to oxygen deprivation and other forms of brain injury. Urgent surgery is often required in the first few weeks of life to improve functioning of the heart, but this surgery also carries a risk of additional brain injuries.

The aim of this study is to provide a better understanding of factors associated with the development of brain injury in neonates undergoing heart surgery in the first year or life. The short-term aim of this study is to provide data to help our team to develop advanced monitoring software that can be used to guide perfusion of the brain during surgery with a view to preventing surgery-related brain injury. The mid-term goal of the study is to identify risk factors associated with brain injury and inflammation around the time of surgery, through using MRI and taking blood samples. A longer term aim of this study is to be able to follow the children as they develop to see if any problems develop later in life. In this study, we will ask parents to complete two brief questionnaires when their infant reaches 2 years of age. Overall, this study aims to improve our understanding of the causes of brain injury in patients born with congenital heart problems. The data provided by this study will help us to develop new tools for monitoring brain perfusion during surgery.

DETAILED DESCRIPTION:
This is a prospective observational exploratory study with the main aim of gathering patient-specific physiological measurements, and early outcome data to support the development of brain neuromonitoring software. We will use this as an opportunity to explore the complex and multi-factorial causes of brain injury and long-term developmental issues in babies undergoing surgery to correct a congenital cardiac condition under one year of age. Demographic, birth, and surgery/PICU risk factors for brain injury identified from a systematic review of previous literature will be recorded. These data will be accompanied by assessment of early post-operative outcomes, intra-operative physiological, blood and neuro monitoring, and assessment of blood and imaging biomarkers.

Specific information recorded or measured as part of this study will include:

Baseline pre-operative procedures:

* Demographic and delivery data will be obtained from the patient's medical records .
* Additional measurement of baseline brain blood flow (Middle Cerebral Artery Cerebral Blood Flow velocity (MCA CBFv)) using Transcranial Doppler (TCD) ultrasound.
* Preoperative brain MRI (obtained without an additional anesthetic or sedation using a feed and swaddle method).
* Blood test; for brain injury and inflammation biomarkers.

Intra-operative measurements

* Operative transcript and relevant surgery information obtained from the patient's notes.
* Routine intraoperative monitoring, including blood analysis, vital signs monitoring, and cerebral oxygenation measurements will be recorded to a laptop for further analysis.
* Continuous measurement of brain blood flow (Middle Cerebral Artery Cerebral Blood Flow velocity (MCA CBFv)) will be performed using Transcranial Doppler (TCD) ultrasound.

Post-operative measurements

* Information reflecting early post-operative outcome will be recorded from the patient's notes.
* Additional measurements of baseline brain blood flow (Middle Cerebral Artery Cerebral Blood Flow velocity (MCA CBFv)) using Transcranial Doppler (TCD) ultrasound will be obtained in the Paediatric Intensive Care Unit.
* Post-operative brain MRI will be obtained without an additional anesthetic or sedation using a feed and swaddle method as soon as the patient is stable and considered well enough to undergo an MRI scan. This decision will be made by the patient's consultant.
* Blood test; for brain injury and inflammation biomarkers.

Cognitive and behavioural follow-up at 2 years:

* Parent-completed Questionnaire (PARCA-R).
* Parent-completed Strengths and Difficulties Questionnaire (SDQ)
* Review of medical notes.

ELIGIBILITY:
Inclusion Criteria:

* Parents/Carers should be willing to provide written informed consent for their child to participate in the study
* Patients should be under 1 year of age.
* Patients with congenital cardiac conditions of any type and severity can be included
* Patients undergo cardiac surgery (any strategy).

Exclusion Criteria:

* Unable (in the investigator's opinion) to comply with the study requirements.
* Known pre-existing brain conditions, and genetic or inflammatory syndromes known to affect brain development.

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Babies (<1 year) undergoing surgery for congenital cardiac disease
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Estimation of brain tissue perfusion and oxygenation. | During paediatric cardiac surgery
  To provide preliminary data to support the development of a prototype intraoperative neuromonitoring system for personalised estimation of brain tissue perfusion and oxygenation during paediatric cardiac surgery.

SECONDARY OUTCOMES:
Identification of modifiable risk factors | Post surgery to 2 years
  Longer-term secondary objectives of the study involve identification of modifiable risk factors associated with post-surgery brain injury and cognitive and behavioural outcomes at 2 years. A predictive statistical model will be developed based on information relating to the patient's brain blood flow management during surgery, as well as demographic factors, such as gestational age and condition at birth, treatment course, and inflammatory and brain injury biomarkers. Outcome data will include pre- and post-surgery brain MRI scans (in a sub-study of 30 patients) and cognitive and behavioural assessment at 2 years of age.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Chung, Principal Investigator — University of Leicester
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No